CLINICAL TRIAL: NCT00692159
Title: Open Label Phase 1 Dose Finding Study of TRC102 in Combination With Pemetrexed in Patients With Advanced or Metastatic Solid Cancer for Whom Curative Therapy is Unavailable
Brief Title: Study of TRC102 in Combination With Pemetrexed in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Bryan Leigh, MD, Medical Monitor, TRACON Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102ST101
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Neoplasm
Keywords: TRC102; Methoxyamine HCL; Pemetrexed; Alimta; Tracon; Phase 1; Cancer; BER; Base Excision Repair; Small Molecule; Anti-folate; Solid Tumor; Neoplastic Processes; Pathologic Processes; Pathological Conditions, Signs and Symptoms
MeSH Terms: conditions — Neoplasms; Neoplastic Processes; Pathologic Processes; Pathological Conditions, Signs and Symptoms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Dose finding single arm
  Interventions: Drug: TRC102 + pemetrexed

INTERVENTIONS:
Drug: TRC102 + pemetrexed — Oral TRC102 solution + IV pemetrexed
  Other Names: Alimta

SUMMARY:
This study is being performed to evaluate the safety and tolerability of TRC102 in combination with Alimta. In addition to safety, this study will also evaluate pharmacokinetics and tumor response.

DETAILED DESCRIPTION:
This study is being performed to evaluate the safety and tolerability of TRC102 in combination with Alimta. In addition to safety, this study will also evaluate pharmacokinetics and tumor response.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given informed consent
* The patient is willing and able to abide by the protocol
* The patient has cancer and curative therapy is unavailable or standard therapy has failed
* The patient is at least 18 years of age
* The patient has adequate ability to perform activities of daily living
* The patient has recovered from significant toxicities of previous therapy
* The patient has adequate organ function as assessed by laboratory testing

Exclusion Criteria:

* The patient has had prior treatment with high-dose chemotherapy requiring stem cell rescue
* The patient is currently on treatment on another therapeutic clinical trial or has received an investigational drug within 4 weeks prior to first dose on this study
* The patient has had prior surgery, radiation or systemic therapy within 4 weeks of starting the study
* The patient has a history of CNS cancer
* The patient has an unstable medical condition including (not limited to) cardiac disease, HIV/AIDS, history of stroke, hepatitis or significant paricardial, pleural or peritoneal effusion
* The patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the recommended Phase 2 dose and overall safety and tolerability of TRC102 when given alone and when combined with pemetrexed for the treatment of patients with advanced solid or metastatic cancer for whom curative therapy is unavailable. | Study completion

SECONDARY OUTCOMES:
Characterize pharmacokinetics, assess anti-tumor activity, and assess pharmacodynamics | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Leigh, MD, Study Director — Tracon Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - Santa Monica, California
  - Cleveland, Ohio

REFERENCES:
- [Derived] Gordon MS, Rosen LS, Mendelson D, Ramanathan RK, Goldman J, Liu L, Xu Y, Gerson SL, Anthony SP, Figg WD, Spencer S, Adams BJ, Theuer CP, Leigh BR, Weiss GJ. A phase 1 study of TRC102, an inhibitor of base excision repair, and pemetrexed in patients with advanced solid tumors. Invest New Drugs. 2013 Jun;31(3):714-23. doi: 10.1007/s10637-012-9876-9. Epub 2012 Sep 29. PMID 23054206
- See also: TRACON Pharmaceuticals Inc. Web Site — http://www.traconpharma.com